CLINICAL TRIAL: NCT03017170
Title: A Randomized, Double-blind, Placebo Controlled Study to Evaluate the Efficacy of Dried Cranberry at 500 mg Daily in Women With Dry Overactive Bladder for 6 Months
Brief Title: Evaluation of the Effect of Dried Cranberry Powder in Women With Dry OAB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Naturex-Dbs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1506016303
Record Dates: First submitted 2016-12-22; First posted 2017-01-11 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cranberry (Experimental): 500mg Dried Cranberry
  Interventions: Drug: Dried Cranberry
- Placebo Oral Capsule (Placebo Comparator): Color Matching Placebo
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Dried Cranberry — Dried cranberry powder is not an "extract" of cranberries, but a "full spectrum" ingredient. It is comprised of a proprietary ratio of dried cranberry fruit, cranberry pomace, and cranberry seeds, each of which is a recognized food and/or dietary ingredient. One 500 mg capsule of dried cranberry powder consists of approximately 25 grams of cranberry fruit.
  Other Names: Cranberry
  Arms: Cranberry
Drug: Placebo Oral Capsule — Colored Maltodextrin: Proprietary mixture of: maltodextrin and food grade colors
  Other Names: Placebo
  Arms: Placebo Oral Capsule

SUMMARY:
A randomized, double-blind, placebo controlled study to evaluate the efficacy of dried cranberry at 500 mg daily in women with overactive bladder for 6-months.

DETAILED DESCRIPTION:
This is a 6 month, randomized, prospective, single-center trial that will be conducted in an outpatient setting at a tertiary care facility. This will be a double-blind, randomized, placebo-controlled parallel study of dried cranberry for OAB symptoms in women. Eligible subjects will be female outpatients aged ≥18 years who have been diagnosed with OAB. All patients will be provided written informed consent before entering the study. The study protocol and all amendments will be approved by the appropriate Institutional Review Board. Patients will be recruited for the study from the office of Dr. Bilal Chughtai, from within Weill Cornell Medical College, including referral by WCMC-affiliated primary care and other physicians not involved with the study, as well as recruited from advertisement (Craigslist, newspapers, posters, etc.). Recruitment will also take place within New York Presbyterian Hospital.

Subjects will have a complete history and physical examination in the office; the participants will complete the validated questionnaires and informed consent, as well as urinalysis. Eligible participants will be enrolled in the study and randomized to receive either a dried cranberry or placebo. The primary endpoint is the mean change in number of voids per day as measured using a three-day voiding diaries from baseline to end-of-treatment. Patients will complete voiding diaries for 3 consecutive days prior to each clinic visit. Secondary endpoints will include a comparison of the patient's baseline OAB symptom bother and quality of life, and sexual function as measured by 4 validated questionnaires: the OABQ-SF, PPBC, SQOL-F, and PFDI-20.

The subjects will be given a device to measure their urinary volume throughout the study.

The study duration will be 6 months. Follow-up visits will be conducted at 12 and 24 weeks. Adverse reactions and complications will be obtained and recorded by Clavien-Dindo Grading System.

The investigator seeks to determine if dried cranberry powder changes the microbiome of women with Overactive Bladder symptoms versus placebo. At visit two (baseline) and visit four (end of study visit) stool and urine samples will be collected from up to 40 study participants out of the 76 participants enrolled in the study. The stool and urine samples will be collected and the microbiome of each specimen will be analyzed by Genomics Core or Epigenomics Core at Weill Cornell Medical College.

Participants in the study will provide urine samples. The urine sample will be collected in sterile containers. Participants in the study will provide one urine sample during visit 2 (Baseline visit) and another sample during visit 4 (end of study). These samples will be subsequently analyzed for the presence/ absence of microbiota. This includes DNA extraction, library preparation, shotgun next-generation sequencing, and follow-up metagenomics and microbiome analysis using bioinformatics alignment tools, in order to identify microbial species and strains. Participants in the study will provide one stool sample during visit 2 of the study and another during visit 4 of the study. Stool samples will be self-collected using a clean catching receptacle (e.g. plastic inverted hat) and plastic scoop to transfer feces into 6 sterile tubes.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory female subject ≥ 18 years of age and able to use the toilet without difficulty
* OAB symptoms for ≥ 6 months
* Frequency of micturition ≥ 8 times per 24 hr and ≥ 3 episodes of urgency (grade 3 or 4) without incontinence during the 3-day micturition diary period at baseline
* Subjects are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study
* Speak English and are able to understand the nature of the study
* Able to give signed written informed consent
* Signed informed consent form

Exclusion Criteria:

* Significant bladder outflow obstruction
* Urinary Incontinence (defined as greater than 3 incontinence episodes in the month prior to screening)
* Catheterization (indwelling catheter)
* Diabetic neuropathy and unstable diabetes mellitus
* Urinary tract infection (UTI) at screening and recurrent UTI defined as ≥ 3 UTIs in the previous 12 months
* Urethral diverticulum
* Neurogenic bladder
* Chronic urologic inflammatory condition (Interstitial cystitis, urethral syndrome, painful bladder syndrome)
* Bladder stones
* History of carcinoma of the urinary tract
* Lower urinary tract surgery in the last 6 months
* Abnormal baseline urinalysis
* Previous pelvic radiation therapy or previous, current malignant disease of the pelvic organs or has received intravesical injection or electrostimluation in the past 12 months
* Planning to undergo urologic procedures for which mucosal bleeding is anticipated
* Drug or Nondrug treatments of OAB (in the previous 56 days), Concomitant medications that affect detrusor activity
* Cerebrovascular diseases
* Neurological impairment or psychiatric disorder preventing appropriate understanding of consent and ability to comply with site personnel instructions
* History of drug or alcohol abuse within the last 12 months.
* Has participated in a study involving the administration of an investigational agent within the past 30 days, or within six half-lives of the prior investigational agent, whichever is longer.
* Subjects on Warfarin
* Females of childbearing potential who are pregnant or planning to become pregnant during the course of the study or breast-feeding
* Subjects with history of kidneys stones
* Treatable condition that could cause urinary incontinence or urgency
* Planning to undergo urologic procedures for which mucosal bleeding is anticipated
* Previous allergic conditions to cranberry products
* Gastrointestinal obstruction or retention or fecal impaction
* Failure to complete baseline 3-day diary
* Subjects unable to swallow the capsule of the intervention
* Subjects with gross hematuria
* Judged by the investigator to be unsuitable for enrollment in this study for any reason
* Allergy or sensitivity to aspirin
* Aspirin dose > 81 mg
* Subjects taking other prescription anti-platelet agents (e.g. clopidogrel, ticlopidine, prasugrel, and ticagrelor)
* Subject has moderate to severe hepatic impairment (Child-Pugh class B or C)
* Subject has severe renal impairment defined as eGFR<30 mL/min/1.73 m2)

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Mean change in number of micturitions per day from baseline until end of treatment | 6 Months

SECONDARY OUTCOMES:
Change in number of urgency and frequency episodes per 24 hours from baseline until end of treatment | 6 Months
Change in number of micturitions occuring during the night from baseline until end of treatment | 6 Months
Change in overactive bladder questionnaire short form (OABQ-SF) score | 6 Months
Change in patient perception of bladder condition (PPBC) score | 6 Months
Change in Sexual Quality of Life-Female (SQOL-F) score | 6 Months
Change in Pelvic Floor Distress Inventory (PFDI-20) | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Chughtai, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No